CLINICAL TRIAL: NCT03027570
Title: The Impact of Incorporating an Exergame Activity Application in a Treatment Regimen for Overweight Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bait Balev Hospital (Other)
Collaborators: University of Haifa (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0067-16-BBL
Record Dates: First submitted 2017-01-04; First posted 2017-01-23 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2016-12

CONDITIONS: Body Mass Index; Blood; Sugar, High; Lipid Disorder; Body Image
Keywords: Exergame; Cellular apps; Smartphone; Overweight; Obesity; Children; Physical activity; Fitness; Motivation; BMI
MeSH Terms: conditions — Hyperglycemia; Lipid Metabolism Disorders; Overweight; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): Five-month program at two centers for the treatment of overweight children.
  Interventions: Behavioral: Control
- Exergame activity_EXG (Experimental): Adding an exergame activity application to the regimen at a center for the treatment of overweight children.
  Interventions: Behavioral: Exergame activity_EXG; Other: Application activity

INTERVENTIONS:
Behavioral: Control — Five-month interdisciplinary program, including: twice a week one-hour group exercise activity sessions, 3-5 group meetings with a dietician, 12-13 parent sessions with a social worker, and a healthy cooking workshop, each child will take part in individual sessions including: two appointments with a pediatrician, three sessions with a dietician and two sessions with a physical therapist serving as a consultant for physical activity.
  Arms: Control
Behavioral: Exergame activity_EXG — In addition to the treatment given to the control group (as described above), the EXG group will obtain home access to the app "Just Dance Now" and part of a weekly exercise session will include a group activity with the app.
  Arms: Exergame activity_EXG
Other: Application activity — The application - "Just Dance Now" will be downloaded to the cellular phone of the child or parent. Exercise using the app will be used by cell phone connection to the child's home computer and as part of exercise group activity.
  Arms: Exergame activity_EXG

SUMMARY:
80 children aged 5-13, BMI≥85%, will be recruited to a program for the treatment of overweight children.The intervention group will use the app "Just Dance Now" and The control group will be exposed to the usual program without the app. Measurements will be performed at the beginning of the program, the end and 3 months after completion of the intervention.

DETAILED DESCRIPTION:
80 children aged 5-13, BMI≥85%, will be recruited to the five-month program, at two centers for the treatment of overweight children. The intervention group will use the app "Just Dance Now" and part of a weekly exercise session will be dedicated to a group app activity. The control group will be exposed to the usual program without the app.

Measurements of BMI, blood sugar and lipid profiles, as well as physical examination, and questionnaires regarding attitude and response to physical activity will be performed at the beginning of the program, the end and 3 months after completion of the intervention. Participation in the sessions will be documented and home activity recorded using a weekly log. ANOVA two-way repeated measures will be used to assess improvements in outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-13 from the center for the treatment of overweight children in the MACABI health organization
* BMI≥85%.

Exclusion Criteria:

* Children with physical disabilities, that don't allow participation in physical activity during the study.
* Children who don't own a mobile phone or don't have an access to a computer to activate the app for one hour a day.
* BMI<85%

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Changes in Body Mass index (BMI) score | 5-8 months

SECONDARY OUTCOMES:
Changes in Behavioral Regulation in Exercise | 5-8 months
  Determined using an Exercise regulation questionnaire (BREQ-2)
Changes in Physical Self-Perception Profile | 5-8 months
  Determined using a Physical Self-Perception Profile questionnaire (PSPP).
Changes in Response toward home physical activity | 5-8 months
  By filling a weekly activity log.
Changes in Response toward physical activity sessions | 5-8 months
  By filling physical activity session attendance.
Changes in Level of physical activity | 5-8 months
  By using a Physical Activity Questionnaire - for elementary School (PAQ-C).
Blood sugar profile | 5-8 months
  By measuring levels of HBAa1c and fasting glucose.
Blood lipid profile | 5-8 months
  By measuring levels of ADL, HDL, and Triglycerides.
Aerobic capacity | 5-8 months
  By using Modified YO-YO IR1 field test to estimate VO2Max levels.
Speed and Agility | 5-8 months
  By using 10*4 - Shuttle Run field test.
Leg endurance ability | 5-8 months
  By using Wall Sit up field test.
Lower limb explosive power | 5-8 months
  By using Standing Long Jump field test.
Forearm muscle strength | 5-8 months
  By using a hand grip failed test.
Coordination levels | 5-8 months
  By using Modified Alternate Hand Wall Toss filed Test

CONTACTS AND LOCATIONS:
Overall Officials: Shai Kremer, MD, Principal Investigator — Maccabi health organization
Locations (1):
- Centers for the treatment of overweight children - MACCABI health organization, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No